CLINICAL TRIAL: NCT07038564
Title: A Clinical Evaluation of the Relationship Between Preoperative Immune-Nutritional Scores and Postoperative Sleep Quality in Women Undergoing Total Abdominal Hysterectomy
Brief Title: Immune-Nutritional Scores and Sleep Quality After Total Abdominal Hysterectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Haseki Training and Research Hospital
Other Study IDs: TAH PNI HALP
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Immune-Nutritional Indexes (PNI, HALP); Postoperative Sleep Quality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Immune-Nutritional Scoring and Postoperative Sleep Assessment — Routine preoperative laboratory data (hemoglobin, albumin, lymphocyte, platelet) will be used to calculate immune-nutritional scores (HALP, PNI). Postoperative sleep quality will be assessed with the Richards-Campbell Sleep Questionnaire (RCSQ).

SUMMARY:
This prospective observational study aims to evaluate the relationship between preoperative immune-nutritional status and postoperative sleep quality in women undergoing total abdominal hysterectomy under general anesthesia. Immune-nutritional scores, including the Prognostic Nutritional Index (PNI) and Hemoglobin-Albumin-Lymphocyte-Platelet (HALP) score, will be calculated using routine preoperative blood parameters. Postoperative sleep quality will be assessed using the Richards-Campbell Sleep Questionnaire (RCSQ). Secondary outcomes include postoperative pain scores and patient satisfaction. The study will enroll 60 patients and seeks to determine whether preoperative physiological markers can predict subjective recovery parameters such as sleep and comfort, potentially contributing to personalized perioperative care.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-70
* ASA physical status I-III
* Undergoing elective total abdominal hysterectomy under general anesthesia
* Available complete blood count and biochemistry results within 24 hours preoperatively
* Planned to stay at least one night postoperatively
* Sufficient cognitive ability to understand and complete questionnaires
* Provided written informed consent

Exclusion Criteria:

* History of neurological or psychiatric illness
* Diagnosed sleep disorders
* Current use of sedative or hypnotic medications
* Undergoing additional surgical procedures during operation
* Requiring postoperative intensive care
* Operated under spinal or epidural anesthesia

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants only. The study population includes women aged 18 to 70 undergoing elective total abdominal hysterectomy under general anesthesia.
Study Population: The study population consists of female patients aged 18 to 70 years undergoing elective total abdominal hysterectomy under general anesthesia at Haseki Training and Research Hospital. Participants must have available preoperative laboratory data and be able to complete postoperative questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Sleep Quality Score | Postoperative first night
  Sleep quality will be measured using the Richards-Campbell Sleep Questionnaire (RCSQ), a validated 5-item instrument assessing sleep depth, latency, number of awakenings, efficiency, and overall quality. Each item is scored from 0 to 100, with higher scores indicating better sleep quality.

SECONDARY OUTCOMES:
Postoperative Pain Score | Post-anesthesia care unit (PACU), postoperative day 1 and day 2 (rest and mobilization)
  Pain levels will be assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst pain imaginable). Scores will be recorded at rest and during mobilization on each postoperative day.
Patient Satisfaction Score | Postoperative day 2
  Overall patient satisfaction with the perioperative experience will be assessed using a 0-10 numeric rating scale, with higher scores indicating greater satisfaction.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li J, Guo Q, Ye X, Lin J, Yi C, Mao H, Yang X, Yu X. Prevalence and risk factors of sleep disturbance in continuous ambulatory peritoneal dialysis patients in Guangzhou, southern China. Int Urol Nephrol. 2012 Jun;44(3):929-36. doi: 10.1007/s11255-011-0060-5. Epub 2011 Sep 30. PMID 21960370
- [Result] Ishiguro T, Aoyama T, Ju M, Kazama K, Fukuda M, Kanai H, Sawazaki S, Tamagawa H, Tamagawa A, Cho H, Hara K, Numata M, Hashimoto I, Maezawa Y, Segami K, Oshima T, Saito A, Yukawa N, Rino Y. Prognostic Nutritional Index as a Predictor of Prognosis in Postoperative Patients With Gastric Cancer. In Vivo. 2023 May-Jun;37(3):1290-1296. doi: 10.21873/invivo.13207. PMID 37103068
- [Result] Farag CM, Antar R, Akosman S, Ng M, Whalen MJ. What is hemoglobin, albumin, lymphocyte, platelet (HALP) score? A comprehensive literature review of HALP's prognostic ability in different cancer types. Oncotarget. 2023 Feb 25;14:153-172. doi: 10.18632/oncotarget.28367. PMID 36848404
- [Result] Para E, Uslu N. Cerrahi hastalarında ameliyat sonrası uyku kalitesi ve uyku düzenini etkileyen etmenler. CBU Sağlık Bilimleri Dergisi. 2022;9(3):443-450. doi:10.34087/cbusbed.1034063.